CLINICAL TRIAL: NCT00004335
Title: Study of Gonadotropin-Releasing Hormone Pulse Frequency in Sexual Maturation and in the Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Michigan (Other)
Other Study IDs: 199/11894; UMMC-271
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Hypogonadism; Precocious Puberty
Keywords: endocrine disorders; growth hormone deficiency; hypogonadism; precocious puberty; rare disease
MeSH Terms: conditions — Hypogonadism; Puberty, Precocious; Endocrine System Diseases; Dwarfism, Pituitary; Rare Diseases

SUMMARY:
OBJECTIVES: I. Evaluate the sleep-entrained patterns of gonadotropin-releasing hormone (GnRH) and sex steroid secretion in normal and hypogonadal children.

II. Examine the acute effects of sex steroids on the sleep-entrained patterns of GnRH secretion in pubertal children and normal adults, either by stimulation of endogenous production with pulsatile injection or by intravenous infusion of GnRH.

III. Examine the role of endogenous opioids by means of opioid receptor blockade in the sex steroid regulation of GnRH secretion in pubertal children and normal adults.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This project involves several clinical protocols that study the regulation and role of pulsatile gonadotropin-releasing hormone (GnRH) secretion.

Studies include dynamic and repeated stimulation tests of pulsatile GnRH; plasma luteinizing hormone, follicular-stimulating hormone, testosterone (T), estradiol (E2), and GnRH measurements at cyclic and episodic intervals; and evaluation of adrenal androgen patterns.

Circadian rhythms of GnRH secretion are monitored during sleep and awake hours. Growth hormone secretory patterns and responses to provocative stimuli are studied as clinically indicated.

Selected participants undergo an assessment of pituitary responsiveness following T, E2, and/or naloxone infusions. The suppressive effects of E2 are also studied during the early follicular phase of the menstrual cycle.

Endocrinologically normal children and normal adult men and women are also studied.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Suspected or proven hypothalamic-pituitary-gonadal dysfunction, i.e.: Significant short stature and possible hypopituitarism Delayed adolescence Precocious puberty Isolated growth hormone deficiency (IGHD)Primary hypogonadism
* Women are also studied, including those with the following disorders: Infertility Oligo- or amenorrhea Hirsutism

--Patient Characteristics--

* Age: 7 to 16 (18 to 35 for women and volunteers)
* Other: No pregnant or nursing women No prisoners Not in neuropsychiatric institute or other facility for mental illness

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 1993-04

CONTACTS AND LOCATIONS:
Overall Officials: Carol M. Foster, Study Chair — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States